CLINICAL TRIAL: NCT04659616
Title: A Multicenter, Phase 1, Open-Label Study of the FGFR Inhibitor Pemigatinib (INCB054828) Administered After Chemotherapy in Newly Diagnosed Acute Myeloid Leukemia (AML) With Adverse or Intermediate Risk Cytogenetics
Brief Title: Pemigatinib After Chemotherapy for the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Incyte Corporation (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Elie Traer, MD PhD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020009; NCI-2020-05267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020009 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-08-20; First posted 2020-12-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Fluid Therapy; Biopsy; Cytarabine; Daunorubicin; pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cytarabine, daunorubicin, pemigatinib) (Experimental): INDUCTION: Patients receive cytarabine IV on days 1-7, daunorubicin IV on days 1-3, and pemigatinib PO QD on days 8-21 in the absence of disease progression or unacceptable toxicity. Patients with hematologic count recovery (assessed between days 25-42) after induction proceed to consolidation therapy. Patients undergo ECHO during screening and as clinically indicated on study. Patients undergo blood sample collection and bone marrow aspirate and biopsy during screening and cycle 11 day 21 on study.
  CONSOLIDATION: Patients receive high dose cytarabine IV BID on days 1, 3, and 5 of each cycle, and pemigatinib PO QD on days 8-21 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression of unacceptable toxicity. Patients undergo ECHO as clinically indicated and blood sample collection and bone marrow biopsy and aspirate at the end of consolidation.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Electrocardiography; Drug: Pemigatinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow biopsy and aspirate
  Other Names: BONE MARROW, LIQUID; Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiratie
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Procedure: Electrocardiography — Undergo ECHO
  Other Names: ECG; EKG
Drug: Pemigatinib — Given PO
  Other Names: INCB054828; Pemazyre

SUMMARY:
This phase I trial identifies the best dose and clinical benefit of giving pemigatinib following standard induction chemotherapy in patients with newly diagnosed acute myeloid leukemia. Pemigatinib selectively inhibits FGFR (fibroblast growth factor receptor) activity, a receptor that may contribute to the growth of leukemia cells. The genetic changes responsible for activating the growth of leukemia cells can be unique to each patient and can change during the course of the disease. Chemotherapy drugs, such as cytarabine and daunorubicin work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose of pemigatinib (INC054828) following standard of care induction chemotherapy.

SECONDARY OBJECTIVES:

I. To assess preliminary efficacy associated with study intervention. II. To assess the safety profile of the study intervention. III. To evaluate time-to- marrow recovery between cycles of pemigatinib.

EXPLORATORY OBJECTIVES:

I. Assess minimal residual disease (MRD) by fluorescent in situ hybridization (FISH), reverse transcriptase-polymerase chain reaction (RT-PCR), and/or next-generation sequencing of acute myeloid leukemia (AML) genetic abnormalities in bone marrow and blood.

II. Quantify FGF2/FGFR immunohistochemical staining of marrow core biopsies and compare to historical controls at various timepoints.

III. Assess ex vivo sensitivity of patient-derived mononuclear cells to pemigatinib with and without FGF2 supplementation.

IV. Evaluate pemigatinib-induced changes in stromal expression using cultured bone marrow samples and compare to historical controls.

V. Evaluate the impact of pemigatinib on the need for intravenous (IV) phosphate replacement after chemotherapy.

OUTLINE: This is a dose-escalation study of pemigatinib followed by a dose-expansion study.

INDUCTION: Patients receive cytarabine IV on days 1-7, daunorubicin IV on days 1-3, and pemigatinib orally (PO) once daily (QD) on days 8-21 in the absence of disease progression or unacceptable toxicity. Patients with hematologic count recovery (assessed between days 25-42) after induction proceed to consolidation therapy. Patients undergo echocardiography (ECHO) during screening and as clinically indicated on study. Patients undergo blood sample collection and bone marrow aspirate and biopsy during screening and cycle 11 day 21 on study.

CONSOLIDATION: Patients receive high dose cytarabine IV twice daily (BID) on days 1, 3, and 5 of each cycle, and pemigatinib PO QD on days 8-21 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression of unacceptable toxicity. Patients undergo ECHO as clinically indicated and blood sample collection and bone marrow biopsy and aspirate at the end of consolidation.

After completion of study treatment, patients are followed up every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* PRE-SCREENING INCLUSION CRITERIA: Ability to understand and the willingness to sign a written informed consent document
* PRE-SCREENING INCLUSION CRITERIA: Age >= 18 years at time of informed consent. Both men and women of all races and ethnic groups will be included
* PRE-SCREENING INCLUSION CRITERIA: Participants must consent to a bone marrow aspirate/biopsy that will be collected prior to start of planned 7+3 induction therapy. Patients with known favorable risk AML (2022 European Leukemia Net [ELN] Guidelines) or FLT3 mutations should not be pre-screened. If the risk category is unknown, then it is okay to pre-screen patients for study. Adverse or intermediate risk needs to be confirmed prior to treatment with pemigatinib (during screening period) as outlined below
* TREATMENT INCLUSION CRITERIA: Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* TREATMENT INCLUSION CRITERIA: For both the dose-determining and dose-expansion cohort, study population is limited to: Newly diagnosed, morphologically documented AML, based on the World Health Organization (WHO) 2008 classification, with wild-type FLT3 and cytogenetics or mutations associated with intermediate or adverse prognostic risk per European Leukemia Net (ELN) guidelines. These include:

  * t(9;11)(p21.3;q23.3); MLLT3-KMT2A
  * Cytogenetic abnormalities not classified as favorable
  * t(6;9)(p23;q34.1); DEK-NUP214
  * t(v;11q23.3); KMT2A rearranged
  * t(9;22)(q34.1;q11.2); BCR-ABL1
  * inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2); GATA2,MECOM(EVI1)
  * -5 or del(5q); -7; -17/abn(17p)
  * Complex karyotype - defined as three or more unrelated chromosome abnormalities in the absence of 1 of the WHO-designated recurring translocations or inversions, that is, t(8;21), inv(16) or t(16;16), t(9;11), t(v;11)(v;q23.3), t(6;9), inv(3) or t(3;3); AML with BCR-ABL1
  * Monosomal karyotype - defined by the presence of 1 single monosomy (excluding loss of X or Y) in association with at least 1 additional monosomy or structural chromosome abnormality (excluding core-binding factor AML)
  * Mutated RUNX1 (without favorable risk cytogenetics/mutations)
  * Mutated BCOR (without favorable risk cytogenetics/mutations)
  * Mutated EZH2 (without favorable risk cytogenetics/mutations)
  * Mutated ASXL1 (without favorable risk cytogenetics/mutations)
  * Mutated SF3B1 (without favorable risk cytogenetics/mutations)
  * Mutated SRSF2 (without favorable risk cytogenetics/mutations)
  * Mutated STAG2 (without favorable risk cytogenetics/mutations)
  * Mutated U2AF1, (without favorable risk cytogenetics/mutations)
  * Mutated ZRSR2 (without favorable risk cytogenetics/mutations)
  * Mutated TP53 (mono- or biallelic) at a variant allele fraction of at least 10%
* TREATMENT INCLUSION CRITERIA: Serum creatinine clearance >= 30 mL/min (as calculated by Cockcroft-Gault formula) (on or by day 8 of induction therapy, prior to starting pemigatinib)
* TREATMENT INCLUSION CRITERIA: Serum phosphate within institutional upper limit of normal (ULN) or can be corrected with supplementation/ phosphate binders to be within institutional ULN (on or by day 8 of induction therapy, prior to starting pemigatinib)
* TREATMENT INCLUSION CRITERIA: Serum electrolytes within institutional ULN: potassium, calcium (total, or corrected for serum albumin in case of hypoalbuminemia) and magnesium. If outside of normal limits, participant will be eligible when electrolytes are corrected (on or by day 8 of induction therapy, prior to starting pemigatinib)
* TREATMENT INCLUSION CRITERIA: Total serum bilirubin =< 3 x ULN (on or by day 8 of induction therapy, prior to starting pemigatinib)
* TREATMENT INCLUSION CRITERIA: Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) =< 3 x ULN (on or by day 8 of induction therapy, prior to starting pemigatinib)
* TREATMENT INCLUSION CRITERIA: Participants must consent to standard of care bone marrow aspirate/biopsies during treatment. Bone marrow biopsies will be obtained prior to study, on day 21 (+/- 3 days, if considered institutional standard of care), after recovery from induction therapy, and at the end of consolidation and/or prior to allogeneic stem cell transplant
* TREATMENT INCLUSION CRITERIA: Female participants of childbearing potential must agree to use effective contraception (2 forms of contraception or abstinence) from the screening visit until 6 months following the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* TREATMENT INCLUSION CRITERIA: Male patients of childbearing potential having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use 2 forms of contraception from the screening visit until 3 months following the last dose of study treatment. The male participant must also refrain from sperm donation from the screening visit until 3 months following the last dose of study treatment

Exclusion Criteria:

* PRE-SCREENING EXCLUSION CRITERIA: Diagnosis of acute promyelocytic leukemia (APL, or AML M3 subtype) per WHO classification
* PRE-SCREENING EXCLUSION CRITERIA: AML with FLT3 mutations that qualify for standard of care treatment with 7+3 and midostaurin (e.g. FLT3 ITD or TKD with allelic ratio > 0.05)
* PRE-SCREENING EXCLUSION CRITERIA: Favorable risk AML: inv(16), t(8;21), NPM1 mutations without FLT3-ITD, or in-frame mutations (mono- or biallelic) affecting the basic leucine zipper region of CEBPA
* PRE-SCREENING EXCLUSION CRITERIA: Any cancer-directed therapy within 2 weeks prior to starting planned 7+3 induction regimen, with the exception of hydroxyurea, which is allowed to control white blood cell count, or empiric all-trans retinoic acid (ATRA) for suspected APL
* PRE-SCREENING EXCLUSION CRITERIA: Prior receipt of a selective FGFR inhibitor
* PRE-SCREENING EXCLUSION CRITERIA: Known liver disease
* PRE-SCREENING EXCLUSION CRITERIA: History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues

  * Except for commonly observed calcifications in soft tissues such as the skin, kidney tendon, or vessels due to injury, disease, or aging in the absence of systemic mineral imbalance)
* PRE-SCREENING EXCLUSION CRITERIA: History of hypovitaminosis D being actively treated with supraphysiologic doses (e.g., 50,000 IU/weekly) to replenish the deficiency. Supraphysiologic doses of vitamin D need to be discontinued prior to starting pemigatinib. Vitamin D supplements are allowed
* PRE-SCREENING EXCLUSION CRITERIA: Untreated human immunodeficiency virus (HIV) or active hepatitis C detectable by PCR, or chronic hepatitis B

  * Individuals positive for hepatitis B core antibody who are receiving intravenous immunoglobulin (IVIg) are eligible if HepB PCR is negative
* PRE-SCREENING EXCLUSION CRITERIA: History of cerebrovascular accident or intracranial hemorrhage within 2 months of enrollment
* PRE-SCREENING EXCLUSION CRITERIA: Unwillingness to receive infusion of blood products
* PRE-SCREENING EXCLUSION CRITERIA: Inability to take oral medication
* PRE-SCREENING EXCLUSION CRITERIA: Gastrointestinal condition/disorders that may raise gastric and/or small intestinal pH that could interfere with absorption, metabolism, or excretion of pemigatinib
* PRE-SCREENING EXCLUSION CRITERIA: Known history and/or current evidence of ectopic mineralization/calcification, including (but not limited to): soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcification
* PRE-SCREENING EXCLUSION CRITERIA: Concurrent active malignancy with expected survival of < 1 year
* PRE-SCREENING EXCLUSION CRITERIA: Active central nervous system involvement with AML
* TREATMENT EXCLUSION CRITERIA: Clinically significant coagulation abnormality (e.g., disseminated intravascular coagulation) that is present on or by day 8 of induction therapy prior to starting pemigatinib
* TREATMENT EXCLUSION CRITERIA: Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from day 1 of planned induction therapy, New York Heart Association class III or IV congestive heart failure, and uncontrolled arrhythmia (participants with pacemaker or with atrial fibrillation and well controlled heart rate are allowed). History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful.

  * A screening QT interval by Fridericia's Correction Formula (QTcF) interval > 480 ms will result in exclusion.
  * For participants with an intraventricular conduction delay (QRS interval > 120 ms), the JTc interval may be used in place of the QTc with approval from Sponsor-Investigator. The JTc must be =< 340 ms if JTc is used in place of the QTc.
* TREATMENT EXCLUSION CRITERIA: Left ventricular ejection fraction (LVEF) by echocardiogram < 45% prior to initiating pemigatinib
* TREATMENT EXCLUSION CRITERIA: Active infection that is not well-controlled by antibacterial or antiviral therapy
* TREATMENT EXCLUSION CRITERIA: Current use of prohibited medications including use of any potent CYP3A4 inducers within 14 days or five half-lives (whichever is longer) before the first dose of study drug.

  * Use of CYP3A4 inhibitors should be avoided but, if medically necessary, is permitted with a dose reduction of study drug
  * Use of moderate CYP3A4 inhibitors are permitted.
  * Based on the low overall bioavailability of topical ketoconazole, there are no restrictions on topical ketoconazole
* TREATMENT EXCLUSION CRITERIA: Current use of prohibited medication
* TREATMENT EXCLUSION CRITERIA: Hypersensitivity to pemigatinib, or its excipients, when administered alone
* TREATMENT EXCLUSION CRITERIA: Current evidence of corneal disorder/keratopathy, including (but not limited to): bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, etc., as confirmed by ophthalmologic examination.
* TREATMENT EXCLUSION CRITERIA: Pregnancy or breastfeeding at the time of enrollment
* TREATMENT EXCLUSION CRITERIA: Any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the participant or compliance with the protocol
* TREATMENT EXCLUSION CRITERIA: Active central nervous system involvement with AML
* TREATMENT EXCLUSION CRITERIA: Patients with FLT mutations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | From cycle 1 day 8, until 14 days after cycle 1 day 28 (up to 42 days)
  Will be summarized using the proportion and exact binomial confidence interval. DLTs will be summarized at each dose level by severity and major organ site according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

SECONDARY OUTCOMES:
Rate of composite complete remission (cCR) | From cycle 1 day 1, until blood cell count recovery after induction (day 25-42)
Duration of remission (DOR) | Date of first response (>= immune complete remission) till date of documented relapse assessed up to 2 years from last dose of study intervention
Event-free survival (EFS) | From cycle 1 day 1, until date of primary refractory disease, progression, relapse, or death from any cause, assessed up to 2 years from last dose of study intervention
Relapse-free survival (RFS) | Date of first response (>= complete remission with incomplete blood count recovery [CRi]), until date of relapse or death from any cause, assessed up to 2 years from last dose of study intervention
Overall survival (OS) | From cycle 1 day 1, until date of death from any cause, assessed up to 2 years from last dose of study intervention
  Estimated with the Kaplan-Meier method.
Incidence of treatment-emergent adverse events (TEAEs) | From cycle 1 day 8, until 90 days after last dose of study intervention
  Will be determined for the safety analysis set (i.e., study participants who receive at least one dose of pemigatinib) and the subset of safety evaluable patients treated at the MTD. The point estimate and 95% confidence interval will be reported. Each toxicity event will be tabulated and summarized by severity and major organ site according to the CTCAE v5.0. Will be evaluated in the dose determining and dose expansion cohorts separately as well as combined.
Incidence of non-treatment related adverse events (AEs) | From cycle 1 day 8, until 90 days after last dose of study intervention
  Will be determined for the safety analysis set (i.e., study participants who receive at least one dose of pemigatinib) and the subset of safety evaluable patients treated at the MTD. The point estimate and 95% confidence interval will be reported. Each toxicity event will be tabulated and summarized by severity and major organ site according to the CTCAE v5.0. Will be evaluated in the dose determining and dose expansion cohorts separately as well as combined
Time-to-marrow recovery | Baseline (cycle 1 day 1), until time of count recovery
  Defined as absolute neutrophil count (ANC) >= 1 x 10^9 /L and platelets >= 100 x 10^9/L.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Traer, MD PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

REFERENCES:
- [Derived] Al-Bazaz M, Forstreuter A, Hammada I, Hille J, Wagner JN, Reinert J, Wehrhahn J, Bokemeyer C, Fiedler W. Acute Lymphoblastic Leukemia Characterized by Rare BCR::FGFR1 Translocation: A Case Report With Literature Review. Case Rep Hematol. 2025 Oct 23;2025:8892036. doi: 10.1155/crh/8892036. eCollection 2025. PMID 41180818